CLINICAL TRIAL: NCT03858855
Title: Inhaled Essential Oil Effect on Common Quality of Life Concerns During Cancer Treatment
Brief Title: Inhaled Essential Oil Effect on Common QOL Concerns During Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Amber Williams, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-18136; NCI-2019-00340 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Gastrointestinal Cancer; Neuroendocrine Carcinoma; Skin Cancer
Keywords: aromatherapy; essential oils; Gastrointestinal Cancer; Neuroendocrine Cancer; Melanoma; skin cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Carcinoma, Neuroendocrine; Skin Neoplasms; Melanoma | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (bergamot essential oil) (Experimental): Patients inhale 7 drops of bergamot essential oil using an essential oil administration bottle TID (morning, midday, and evening) for up to 7 days. Patients also use a journal to document symptoms, time of inhalation, and medication use TID for up to 7 days.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Subject Diary
- Group II (chamomile essential oil) (Experimental): Patients inhale 7 drops of chamomile essential oil and complete journal as in group I.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Subject Diary
- Group III (ginger essential oil) (Experimental): Patients inhale 7 drops of ginger essential oil and complete journal as in group I.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Subject Diary
- Group IV (almond essential oil) (Active Comparator): Patients inhale 7 drops of almond essential oil and complete journal as in group I.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Subject Diary

INTERVENTIONS:
Procedure: Aromatherapy and Essential Oils — Use bergamot essential oil
  Other Names: Aromatherapy
  Arms: Group I (bergamot essential oil)
Procedure: Aromatherapy and Essential Oils — Use chamomile essential oil
  Other Names: Aromatherapy
  Arms: Group II (chamomile essential oil)
Procedure: Aromatherapy and Essential Oils — Use ginger essential oil
  Other Names: Aromatherapy
  Arms: Group III (ginger essential oil)
Procedure: Aromatherapy and Essential Oils — Use almond essential oil
  Other Names: Aromatherapy
  Arms: Group IV (almond essential oil)
Other: Subject Diary — Complete journal
  Other Names: Patient Diary; Subj Diary Form; Subject Diary Form

SUMMARY:
This single-blind, randomized controlled trial studies how well inhaled essential oils work for common quality of life concerns in patients who are undergoing cancer treatment such as chemotherapy, targeted therapy, and/or immunotherapy given through the vein (intravenously). Aromatherapy using essential oils, such as ginger essential oil, German chamomile essential oil, and bergamot essential oil, may improve quality of life issues such as nausea, anxiety, loss of appetite, and fatigue in patients undergoing treatment for cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if aromatherapy, specifically inhaled essential oil, is beneficial for side effects related to cancer treatments involving chemotherapy, targeted therapy, and/or immunotherapy administered intravenously.

II. To describe the effect of inhaled ginger essential oil, German chamomile essential oil, and bergamot essential oil on nausea and anxiety of patients receiving chemotherapy, targeted therapy, and/or immunotherapy administered intravenously.

III. To describe the effect of decreased levels of nausea and/or anxiety on levels of appetite and/or fatigue.

IV. To evaluate the acceptability of using a personal inhalation bottle for inhalation of essential oils.

OUTLINE: Patients are randomized to 1 of 4 groups.

GROUP I: Patients inhale 7 drops of bergamot essential oil using a personalized inhalation bottle three times daily (TID) (morning, midday, and evening) for up to 7 days. Patients also use a journal to document symptoms, time of inhalation, and medication use TID for up to 7 days.

GROUP II: Patients inhale 7 drops of chamomile essential oil and complete journal as in group I.

GROUP III: Patients inhale 7 drops of ginger essential oil and complete journal as in group I.

GROUP IV (CONTROL): Patients inhale 7 drops of almond essential oil and complete journal as in group I.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal cancers, neuroendocrine cancer, or melanoma or other skin cancers
* Receiving chemotherapy, targeted therapy, and/or immunotherapy
* Not naive to the treatment
* Must be able to read and write English

Exclusion Criteria:

* Allergies to ragweed, chrysanthemum, chamomile, ginger, bergamot, citrus fruits, tree nuts, perfumes
* Asthma diagnosis
* Patients receiving only octreotide injections
* Patients receiving floxuridine (FUDR) via hepatic artery infusion (HAI) pump only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Effects of essential oils on nausea and anxiety | Up to 7 days
  Levels of nausea and anxiety will be measured using a numerical grading scale of 0-10. 0 will equal "good" meaning no nausea or anxiety. 10 will equal "horrible" meaning the worst nausea or anxiety. Data for each outcome will be collected 3 times a day, for a total of 21 measurements from each subject. For data analysis, we will compress the 21 measures into 3 scores. Each subject will be given a daily outcome level by averaging the 3 measures. The 7 daily outcome levels will become 3 scores by averaging data from days 1 and 2 (Period 1), days 3 and 4 (Period 2), and days 5, 6, and 7 (Period 3). Using the 3 scores, each outcome will be modeled using a repeated measures regression allowing the variability of outcome scores to vary with period. Period, group membership, the interaction between period and group membership, gender, age, and type of cancer will be model predictors. For each outcome, the contrast of interest will be that between each treatment group and the control group.

SECONDARY OUTCOMES:
Determine if decreased levels of nausea and/or anxiety effect appetite and/or fatigue | Up to 7 days
  Anticipated results of the study are that patients will report decreased levels of nausea and anxiety. With the decreased levels of nausea and anxiety, we anticipate that patients will report increased levels of appetite and decreased levels of fatigue. Loss of appetite and fatigue will be measured using a numerical grading scale of 0-10. 0 will equal "good" meaning no loss of appetite or fatigue. 10 will equal "horrible" meaning the worst appetite loss or fatigue. Data will be collected, measured, and analyzed in the same manner as Outcome 1.
Acceptability of using a personal inhalation bottle for inhalation of essential oils - ease of use | Up to 7 days
  The overall ease of using the personal inhalation bottle will be measured through post-study ratings by participants. A numerical rating scale of 1-5 will be used. 1 will equal strongly disagree; 2 will equal disagree; 3 will equal neither agree nor disagree; 4 will equal agree; and 5 will equal strongly agree. The study will compare via a percentage those participants with positive acceptability when compared to those with negative acceptability.
Acceptability of using a personal inhalation bottle for inhalation of essential oils - utilization post study period | Up to 7 days
  The utilization of the personal inhalation bottle beyond the study period will be measured through post-study ratings by participants. A numerical rating scale of 1-5 will be used. 1 will equal strongly disagree; 2 will equal disagree; 3 will equal neither agree nor disagree; 4 will equal agree; and 5 will equal strongly agree. The study will compare via a percentage those participants with positive acceptability when compared to those with negative acceptability.
Acceptability of using a personal inhalation bottle for inhalation of essential oils - perception of benefit of essential oil for symptoms | Up to 7 days
  The overall perception of help for symptoms will be measured through post-study ratings by participants. A numerical rating scale of 1-5 will be used. 1 will equal strongly disagree; 2 will equal disagree; 3 will equal neither agree nor disagree; 4 will equal agree; and 5 will equal strongly agree. The study will compare via a percentage those participants with positive acceptability when compared to those with negative acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Amber Williams, MSN, RN, OCN, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu